CLINICAL TRIAL: NCT01854398
Title: The Effect of Continuous Positive Airway Pressure on Diastolic Function in Patients With Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1-2013-0021
Record Dates: First submitted 2013-05-10; First posted 2013-05-15 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive sleep apnea; Continuous positive airway pressure; diastolic function
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CPAP group (Experimental)
  Interventions: Device: CPAP group
- sham-CPAP group (Sham Comparator)
  Interventions: Device: sham-CPAP group

INTERVENTIONS:
Device: CPAP group — Enrolled patients are randomized to CPAP group or sham-CPAP group by 1:1 ratio. The patients in each group will undergo CPAP or sham-CPAP for 3 months.
  Arms: CPAP group
Device: sham-CPAP group — Enrolled patients are randomized to CPAP group or sham-CPAP group by 1:1 ratio. The patients in each group will undergo CPAP or sham-CPAP for 3 months. Sham CPAP consists of a CPAP machine that is modified to include a large hidden leak in the exhaust port of the mask to disperse the therapeutic pressure.
  Arms: sham-CPAP group

SUMMARY:
The association of obstructive sleep apnea (OSA) and cardiac diastolic dysfunction have been reported, and improvement of diastolic function after continuous positive airway pressure (CPAP) in OSA patients was observed. However, more detailed analysis of diastolic function by supine bicycle exercise echocardiography is lacking. The investigators hypothesized that 3 months of CPAP therapy in OSA patients will significantly improve diastolic functional parameters measured by exercise stress echocardiography. Patients with severe OSA (Apnea-hypopnea index > 30) will be included in this study, and randomized to CPAP versus sham-CPAP group by 1:1 ratio. Supine bicycle exercise echocardiography, pulse wave velocity, 24 hours ambulatory blood pressure (BP), central BP will be checked before and after CPAP therapy and parameters will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Patietns≥20 and ≤75 years-old
* Patients who diagnosed as obstructive sleep apnea and AHI>30 on polysomnography

Exclusion Criteria:

* Age < 20 years-old
* Left ventricular dysfunction (LVEF<50%) or structural heart disease on transthoracic echocardiography
* Diabetes mellitus
* Significant cardiac valvular disease (≥moderate)
* Severe hypertension (>180/110mmHg)
* Moderate or severe kidney disease (eGFR < 60 mL/min )
* Clinically significant liver disease
* History of coronary artery disease
* malignancy or autoimmune disease
* Acute/chronic infection status
* Pregnant status
* Patients taking anxiolytics or sedatives

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-05; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
The differences of supine bicycle exercise echocardiographic parameters and PWV before and after CPAP therapy, and between CPAP group and sham CPAP group. | after 3 months intervention (CPAP)
  The differences of supine bicycle exercise echocardiogrphic parameters (diastolic function grade, mitral inflow parameters, mitral tissue doppler parameters, E/E') and PWV before and after CPAP therapy, and between CPAP group and sham CPAP group.

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Yonsei Cardiovascular Hospital, Yonsei University College of Medicine, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Shim CY, Kim D, Park S, Lee CJ, Cho HJ, Ha JW, Cho YJ, Hong GR. Effects of continuous positive airway pressure therapy on left ventricular diastolic function: a randomised, sham-controlled clinical trial. Eur Respir J. 2018 Jan 31;51(2):1701774. doi: 10.1183/13993003.01774-2017. Print 2018 Feb. PMID 29386335